CLINICAL TRIAL: NCT04211298
Title: Dexmedetomidine Versus Propofol Sedation in Flexible Bronchoscopy: A Randomized Controlled Trial
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Mordechai Kremer, Head of the pulmonary division, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0312-19-RMC
Record Dates: First submitted 2019-12-24; First posted 2019-12-26 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Sedation Complication
MeSH Terms: interventions — Dexmedetomidine; Propofol

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dexmedetomidine (Active Comparator): Dexmedetomidine will be used for sedation during bronchoscopy
  Interventions: Drug: Dexmedetomidine
- Propofol (Placebo Comparator): Propofol will be used for sedation during bronchoscopy
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine will be used for sedation during bronchoscopy
  Arms: Dexmedetomidine
Drug: Propofol — Propofol
  Arms: Propofol

SUMMARY:
The study will evaluate clinical outcomes during bronchoscopy procedures with dexmedetomidine in comparison to propofol.

The clinical outcomes that will be evaluated are: oxygen saturation, transcutaneous Pco2, blood pressure and complications

ELIGIBILITY:
Inclusion Criteria:

* All patients in the age group 18 to 70 years requiring flexible bronchoscopic evaluation of the airway in the Pulmonary institute at Rabin medical center

Exclusion Criteria:

* known or suspected allergy to any of the study drugs, seizure disorder, renal (with serum creatinine > 2 mg/dL) or hepatic impairment (elevated liver enzymes > 2 times normal), haemodynamic instability (bradycardia with HR < 50 bpm or hypotension with SBP < 90 mmHg), or seriously ill patients with American Society of Anesthesiologists' physical status above III

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-05-30 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
number of de-saturation events | During the procedure
  Number of events during bronchoscopy when saturation level decreased under 90%
Oxygen saturation time < 90% | During the procedure
  Total time during the procedure that the oxygen saturation was under 90%

CONTACTS AND LOCATIONS:
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pertzov B, Krasulya B, Azem K, Shostak Y, Izhakian S, Rosengarten D, Kharchenko S, Kramer MR. Dexmedetomidine versus propofol sedation in flexible bronchoscopy: a randomized controlled trial. BMC Pulm Med. 2022 Mar 15;22(1):87. doi: 10.1186/s12890-022-01880-9. PMID 35291989